CLINICAL TRIAL: NCT02600923
Title: STUDY OF PALBOCICLIB IN COMBINATION WITH LETROZOLE AS TREATMENT OF POSTMENOPAUSAL WOMEN WITH HORMONE RECEPTOR POSITIVE, HER2-NEGATIVE ADVANCED BREAST CANCER FOR WHOM LETROZOLE THERAPY IS DEEMED APPROPRIATE
Brief Title: Palbociclib Plus Letrozole For Postmenopausal Women With HR(+) HER2(-) Advanced Breast Cancer For Whom Letrozole Is Deemed Appropriate
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Masking: None | Purpose: Treatment
Other Study IDs: A5481053
Record Dates: First submitted 2015-11-06; First posted 2015-11-09 (Estimated); Results first posted 2020-05-21 (Actual); Last update posted 2022-01-20 (Actual); Status verified 2022-01

CONDITIONS: Advanced Breast Cancer Female
Keywords: palbociclib, ibrance, breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — palbociclib; Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Palbociclib + Letrozole (Experimental): palbociclib and letrozole combination
  Interventions: Drug: Palbociclib; Drug: Letrozole

INTERVENTIONS:
Drug: Palbociclib — Palbociclib will be administered orally once a day at 125 mg/day for 21 days followed by 7 days off treatment for each 28-day cycle (Schedule 3/1).
  Other Names: Ibrance
Drug: Letrozole — Letrozole will be administered orally at 2.5 mg once daily as continuous daily dosing schedule according to product labeling and in compliance with its local prescribing information.
  Other Names: Femara

SUMMARY:
The purpose of this study is to provide access to palbociclib in Mexico and in selected Latin American countries before it becomes commercially available to patients with HR positive/HER2-negative ABC who are appropriate candidates for letrozole therapy.

ELIGIBILITY:
Inclusion Criteria:

* Adult women with proven diagnosis of advanced adenocarcinoma of the breast (locoregional recurrent or metastatic disease).
* Women who are not of childbearing potential.
* ER-positive and/or Progesterone receptor (PgR)-positive tumor based on local laboratory results (test as per local practice).
* HER2-negative breast cancer based on local laboratory results (test as per local practice or local guidelines).
* Patients must be appropriate candidates for letrozole therapy.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
* Adequate bone marrow function.
* Adequate liver function
* Adequate renal function.

Exclusion Criteria:

* Known hypersensitivity to letrozole, or any of its excipients, or to any palbociclib excipients.
* Current use of food or drugs known to be potent inhibitors or inducers of CYP3A4 isoenzymes within 7 days prior to study entry.
* Prior treatment with any CDK inhibitor.
* Previous participation in a palbociclib clinical study.
* Participation in other studies involving investigational drug(s) within 2 weeks prior to study entry and/or during study participation.
* QTc >480 msec; history of QT syndrome, Brugada syndrome or known history of QTc prolongation, or Torsade de Pointes.
* High cardiovascular risk, including, but not limited to recent myocardial infarction, severe/unstable angina and severe cardiac dysrhythmias in the past 6 months prior to enrollment.
* Diagnosis of any second invasive malignancy within the last 3 years prior to enrollment. Note: patients with adequately treated basal cell or squamous cell skin cancer, a history of intraepithelial neoplasia or in situ disease (eg, carcinoma in situ of the cervix or melanoma in situ) may enter.
* Active uncontrolled or symptomatic brain metastases. Previously treated and clinically stable, brain metastases are permitted.
* Other severe acute or chronic medical or psychiatric conditions.
* Patients who are investigational site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the investigator, or patients who are Pfizer employees directly involved in the conduct of the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 131 (Actual)
Dates: Start 2016-04-15 (Actual); Primary Completion 2019-05-28 (Actual); Study Completion 2019-05-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (24):
- Argentina (7):
  - Instituto de Oncologia de Rosario, Rosario, Santa Fe Province
  - Sanatorio Guemes, CABA
  - Hospital Italiano de Buenos Aires, CABA
  - Hospital Britanico de Buenos Aires, CABA
  - Instituto Medico Especializado Alexander Fleming, CABA
  - Instituto de Cardiologia y Cirugia Cardiovascular, Santa Fe
  - ISIS Centro Especializado, Santa Fe
- Brazil (6):
  - Hospital Da Cidade De Passo Fundo, Passo Fundo, Rio Grande do Sul
  - Hospital Sao Lucas da PUCRS / Uniao Brasileira de Educacao e Assistencia, Porto Alegre, Rio Grande do Sul
  - Oncologia Rede D'Or S.A., Rio de Janeiro
  - IDOR - Instituto D'Or em Pesquisa e Ensino, Rio de Janeiro
  - Sociedade Beneficente de Senhoras Hospital Sirio Libanes, São Paulo
  - Clínica de Pesquisa e Centro de Estudos em Oncologia Ginecológica e Mamária Ltda, São Paulo
- Colombia (6):
  - Instituto de Cancerologia S.A., Medellín, Antioquia
  - Administradora Country, Bogotá, Bogota D.C.
  - Oncology Center, Bogotá, Bogota D.C.
  - Oncomedica S.A., Montería, Departamento de Córdoba
  - Imagenes Diagnosticas, Pereira, Risaralda Department
  - ONCOLOGOS DEL OCCIDENTE S.A.S Sede Pereira Clinica de Alta Tecnologia Maraya, Pereira, Risaralda Department
- Mexico (5):
  - Fucam A.C., Coyoacán, D.F.
  - Instituto Nacional de Cancerologia, Tlalpan, D.F.
  - Hospital Maria Auxiliadora, Guadalajara, Jalisco
  - Clinica de Especialidades Medicas Intepro, ONCE Oncologia Especializada, Zapopan, Jalisco
  - Hospital Universitario Dr. Jose Eleuterio Gonzalez, Monterrey, Nuevo León

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Fein L, Lazaretti N, Chuken YL, Benfield JRGR, Mano MS, Lobaton J, Korbenfeld E, Damian F, Lu DR, Mori A, Patyna SJ, Franco S. Expanded Access Study of Palbociclib Plus Letrozole for Postmenopausal Women with HR+/HER2- Advanced Breast Cancer in Latin America for Whom Letrozole Therapy is Deemed Appropriate. Clin Drug Investig. 2023 Sep;43(9):699-706. doi: 10.1007/s40261-023-01294-3. Epub 2023 Aug 18. PMID 37594640
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A5481053

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 131 participants were enrolled and assigned to study treatment, and 130 participants were treated in the study.
Groups:
- Palbociclib+Letrozole: Participants received palbociclib orally once daily at 125 mg for 21 days followed by 7 days off treatment for each 28-day cycle, and letrozole orally at 2.5 mg QD as a continuous daily dosing schedule. Participants continued to receive treatments with palbociclib+letrozole until disease progression, symptomatic deterioration, unacceptable toxicity, death, withdrawal of consent, or time of commercial availability of palbociclib, whichever occurred first.
Period: Overall Study
Arm/Group | Palbociclib+Letrozole
Started | 131
Treated | 130
Completed | 0
Not Completed | 131
Not completed — Death | 10
Not completed — Adverse Event | 3
Not completed — Global deterioration of health status | 2
Not completed — Insufficient clinical response | 6
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 5
Not completed — Objective progression or relapse | 50
Not completed — Study terminated by Sponsor | 53
Not completed — Not treated | 1

BASELINE CHARACTERISTICS:
Population: Baseline analysis population included all participants who received at least 1 dose of palbociclib treatment.
Arm/Group | Palbociclib+Letrozole
Number analyzed (Participants) | 130
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 89
  >=65 years | 41
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 130
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 130
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With All-causality Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a clinical investigation participant administered a product; the event did not need to have a causal relationship with the treatment. All AEs reported after initiation of study drug treatment were considered as TEAE. AE severity was graded according to Common Terminology Criteria for AEs (CTCAE) version 4.03. Grade 1 AEs are mild AEs; Grade 2 AEs are moderate AEs; Grade 3 AEs are severe AEs, Grade 4 AEs are life-threatening consequences and Grade 5 AEs are deaths related to AEs. Each AE was counted once for the participant in the most severe severity.
Time Frame: 3 years
Population: The analysis population included all participants who received at least 1 dose of palbociclib treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Palbociclib+Letrozole
Number analyzed (Participants) | 130
Participants
  Grade 1 | 0
  Grade 2 | 17
  Grade 3 | 82
  Grade 4 | 23
  Grade 5 | 7

2. Primary Outcome: Number of Participants With Palbociclib-related TEAEs
Description: An AE was any untoward medical occurrence in a clinical investigation participant administered a product; the event did not need to have a causal relationship with the treatment. All AEs reported after initiation of study drug treatment were considered as TEAE. AE severity was graded according to CTCAE version 4.03. Grade 1 AEs are mild AEs; Grade 2 AEs are moderate AEs; Grade 3 AEs are severe AEs, Grade 4 AEs are life-threatening consequences and Grade 5 AEs are deaths related to AEs. Palbociclib-related TEAEs were determined by the investigator.
Time Frame: 3 years
Population: The analysis population included all participants who received at least 1 dose of palbociclib treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Palbociclib+Letrozole
Number analyzed (Participants) | 130
Participants
  Grade 1 | 2
  Grade 2 | 25
  Grade 3 | 81
  Grade 4 | 20
  Grade 5 | 0

3. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: An SAE was any untoward medical occurrence at any dose that resulted in death; was life threatening; required inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability/incapacity; resulted in congenital anomaly/birth defect. AEs included both SAEs and AEs. Palbociclib-related SAEs were determined by the investigator.
Time Frame: 3 years
Population: The analysis population included all participants who received at least 1 dose of palbociclib treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Palbociclib+Letrozole
Number analyzed (Participants) | 130
Participants
  All-causality | 32
  Palbociclib-related | 6

4. Secondary Outcome: Number of Participants With Death
Description: Death from any cause while on treatment and within 28 days of palbociclib discontinuation was only counted below.
Time Frame: 3 years
Population: The analysis population included all participants who received at least 1 dose of palbociclib treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Palbociclib+Letrozole
Number analyzed (Participants) | 130
Participants | 5

5. Secondary Outcome: The Objective Response Rate (ORR)
Description: The tumor response was based on the response reported by investigator per local practice. No response confirmation was applied. ORR was defined as the percentage of participants with complete response or partial response relative to all as-treated population.
Time Frame: 3 years
Population: The analysis population included participants with efficacy data contributing to the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of evaluable participants
Arm/Group | Palbociclib+Letrozole
Number analyzed (Participants) | 129
percentage of evaluable participants | 24.8 [17.6 to 33.2]

ADVERSE EVENTS:
Time Frame: 3 years
Description: The same event may appear as both an AE and an SAE. However, what is presented are distinct events. An event may be categorized as serious in 1 participant and as non-serious in another participant, or 1 participant may have experienced both a serious and non-serious event during the study. Total number at risk below refers to the number of participants evaluable for SAEs or AEs.
Arm/Group | Palbociclib+Letrozole
All-Cause Mortality (participants affected / at risk) | 10/130
Serious Adverse Events (participants affected / at risk) | 32/130
Other Adverse Events (participants affected / at risk) | 129/130
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Palbociclib+Letrozole (N=130)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (2)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Disease progression (General disorders) | 2 (2)
General physical health deterioration (General disorders) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Device related infection (Infections and infestations) | 1 (1)
Herpes virus infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 3 (3)
Tuberculosis (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 2 (2)
Fractured ischium (Injury, poisoning and procedural complications) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Tumour flare (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Haemorrhagic stroke (Nervous system disorders) | 1 (1)
Hypertensive hydrocephalus (Nervous system disorders) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 1 (1)
Spinal cord compression (Nervous system disorders) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 2 (3)
Vena cava thrombosis (Vascular disorders) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Palbociclib+Letrozole (N=130)
Anaemia (Blood and lymphatic system disorders) | 44 (111)
Leukopenia (Blood and lymphatic system disorders) | 45 (173)
Lymphopenia (Blood and lymphatic system disorders) | 11 (19)
Neutropenia (Blood and lymphatic system disorders) | 91 (709)
Thrombocytopenia (Blood and lymphatic system disorders) | 32 (89)
Abdominal distension (Gastrointestinal disorders) | 14 (21)
Abdominal pain (Gastrointestinal disorders) | 12 (17)
Abdominal pain upper (Gastrointestinal disorders) | 8 (8)
Constipation (Gastrointestinal disorders) | 21 (24)
Diarrhoea (Gastrointestinal disorders) | 30 (50)
Dyspepsia (Gastrointestinal disorders) | 9 (10)
Nausea (Gastrointestinal disorders) | 25 (34)
Stomatitis (Gastrointestinal disorders) | 8 (15)
Vomiting (Gastrointestinal disorders) | 17 (40)
Asthenia (General disorders) | 22 (33)
Fatigue (General disorders) | 20 (26)
Mucosal inflammation (General disorders) | 11 (26)
Oedema peripheral (General disorders) | 9 (12)
Pyrexia (General disorders) | 8 (9)
Influenza (Infections and infestations) | 10 (11)
Nasopharyngitis (Infections and infestations) | 7 (14)
Upper respiratory tract infection (Infections and infestations) | 15 (21)
Urinary tract infection (Infections and infestations) | 7 (8)
Lymphocyte count decreased (Investigations) | 16 (62)
Neutrophil count decreased (Investigations) | 36 (259)
Platelet count decreased (Investigations) | 19 (50)
White blood cell count decreased (Investigations) | 23 (129)
Decreased appetite (Metabolism and nutrition disorders) | 10 (10)
Arthralgia (Musculoskeletal and connective tissue disorders) | 26 (31)
Back pain (Musculoskeletal and connective tissue disorders) | 21 (33)
Myalgia (Musculoskeletal and connective tissue disorders) | 8 (10)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 15 (23)
Dizziness (Nervous system disorders) | 12 (14)
Headache (Nervous system disorders) | 25 (37)
Insomnia (Psychiatric disorders) | 9 (9)
Cough (Respiratory, thoracic and mediastinal disorders) | 21 (25)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 (10)
Alopecia (Skin and subcutaneous tissue disorders) | 18 (22)
Dry skin (Skin and subcutaneous tissue disorders) | 10 (10)
Pruritus (Skin and subcutaneous tissue disorders) | 7 (7)
Rash (Skin and subcutaneous tissue disorders) | 10 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2015-07-23): https://cdn.clinicaltrials.gov/large-docs/23/NCT02600923/Prot_000.pdf
  • Statistical Analysis Plan (2016-02-04): https://cdn.clinicaltrials.gov/large-docs/23/NCT02600923/SAP_001.pdf